CLINICAL TRIAL: NCT03294928
Title: Arterial Waveform Analysis Applying Different Positive End-Expiratory Pressure (PEEP) Levels in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Prof. Carlo Palombo, Professor, University of Pisa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UPisa - 2017
Record Dates: First submitted 2017-09-19; First posted 2017-09-27 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Blood Pressure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- progressive increasing of PEEP level (Experimental): four-step measurements of central artery blood pressure evaluating contour wave analysis during a progressive increasing of PEEP level.
  Interventions: Other: progressive increasing of PEEP level.

INTERVENTIONS:
Other: progressive increasing of PEEP level. — four-step measurements of central artery blood pressure evaluating contour wave analysis during a progressive increasing of PEEP level First step (Baseline) Subjects spontaneously breathe in air at atmospheric pressure during applanation tonometry.
  Second step (PEEP=5 cm H2O) Applanation tonometry was performed during the application of PEEP = 5 cmH2O (Oxygen flow = 8lt.- Air flow = 10 lt.).
  Third step (PEEP= 10 cm H2O) Applanation tonometry was performed during the application of PEEP = 10 cmH2O (Oxygen flow = 15lt.- Air flow = 20 lt.).
  Fourth step (Recovery) Subjects spontaneously rebreathe air at atmospheric pressure during applanation tonometry.

SUMMARY:
Population in study will be selected from students and staff of the University of Pisa. Right carotid artery contour wave analysis will be performed during the application of different PEEP levels (from 0 cmH2O to 10 cmH2O) with applanation tonometry technique.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 40, absence of any chronic diseases, no smoke, no drugs assumptions, no use of caffeine the day of the exam

Exclusion Criteria:

* pregnancy, chronic diseases, smokers, and intake of caffeine the day of the exam.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2017-10-05 (Actual); Study Completion 2017-10-15 (Actual)

PRIMARY OUTCOMES:
hemodynamic variations in wave reflection induced by the application of increasing levels of PEEP in healthy subjects. | at rest and after 5 minutes
  Mean blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pisa, Pisa, Italy

REFERENCES:
- [Derived] Belfiore J, Brogi E, Nicolini N, Deffenu D, Forfori F, Palombo C. Hemodynamic variations in arterial wave reflection associated with the application of increasing levels of PEEP in healthy subjects. Sci Rep. 2022 Feb 28;12(1):3335. doi: 10.1038/s41598-022-07410-1. PMID 35228629